CLINICAL TRIAL: NCT03714022
Title: A Randomized, Open-Label, Parallel-Group, Single-dose, Biocomparability Study of the Pharmacokinetics of the Abatacept (BMS-188667) Drug Product Converted From Drug Substance of a New Abatacept Drug Substance Process Relative to the Current Abatacept Drug Process in Healthy Participants
Brief Title: A Study to Evaluate the Pharmacokinetics of Abatacept Converted From Drug Substance by Two Different Processes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-682
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive abatacept at a single dose of 750 mg as IV infusion on Day 1 converted from drug substance by a new process.
  Interventions: Drug: Abatacept
- Treatment B (Active Comparator): Participants will receive abatacept at a single dose 750 mg as IV infusion on Day 1 converted from drug substance by converted from drug substance by the current process.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Participants will receive abatacept at a single dose 750 mg as IV infusion.

SUMMARY:
The main objective of this study is to compare the pharmacokinetics (PK) of the abatacept drug product converted from drug substance by a new drug substance process (Treatment A) relative to the current drug substance process (Treatment B) following a single dose (750 mg) intravenous (IV) infusion in healthy participants.

DETAILED DESCRIPTION:
Participants will be admitted to the clinical facility the day prior to dosing (Day -1) and will be confined until at least 24 hours post-dose. On Day 1, eligible participants will be randomized in a 1:1 ratio to either Treatment A or Treatment B. The randomization will be stratified by weight categories: >= 60 to < 70 kg, >= 70 to < 80 kg, >= 80 to < 90 kg, and >= 90 to <= 100 kg.

ELIGIBILITY:
Inclusion Criteria:

* Body weight will be between 60 and 100 kg, inclusive.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 24 hours prior to the start of study treatment.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with abatacept plus 5 half-lives of abatacept (85 days) plus 30 days (duration of ovulatory cycle) for a total of 115 days post-treatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with abatacept plus 5 half-lives of abatacept (85 days) plus the duration of spermatogenesis (90 days) for a total of 175 days after the last dose of study treatment. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Participants who have a present malignancy or previous malignancy within the last 5 years prior to screening (except documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ). Participants who had a screening procedure that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations.
* Participants with a history of herpes zoster.
* Donation of blood to a blood bank or in a clinical study (except a screening visit or follow-up visit) within 4 weeks of study treatment administration (within 2 weeks of study treatment administration for plasma only).
* Blood transfusion within 4 weeks of study treatment administration.
* Recent (within 6 months of study treatment administration) history of smoking or current smokers. This includes participants using electronic cigarettes or nicotine-containing products such as tobacco for chewing, nicotine patches, nicotine lozenges, or nicotine gum.
* History of allergy to abatacept or related compounds.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Qps-Mra, Llc, South Miami, Florida
  - PPD Development, LP, Austin, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 140 participants were randomized and treated.
Groups:
- Cohort A (New Process): Participants received a single IV infusion (750 mg) of Abatacept drug product converted from drug substance by a new process
- Cohort B (Current Process): Participants received a single IV infusion (750 mg) of Abatacept drug product converted from drug substance by the current process
Period: Overall Study
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Started | 70 | 70
Completed | 66 | 67
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Consent withdrawal | 0 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (New Process) | Cohort B (Current Process) | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.4 (9.29) | 36.6 (9.37) | 36.5 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 41 | 44 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 44 | 84
  Not Hispanic or Latino | 30 | 26 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 29 | 51
  White | 45 | 39 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Maximum Observed Serum Concentration
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
ug/mL | 237.0341 (26) | 236.2882 (23)
Statistical Analysis 1: Comparison: Cohort A (New Process) vs Cohort B (Current Process); Test type: Equivalence — Equivalence is concluded if the 90% CIs for the ratios of geometric means are contained within 0.8 to 1.25; Ratio of Geometric Means = 0.998, 90% CI 2-sided [0.941 to 1.058] — Cohort A vs Cohort B

2. Primary Outcome: Area Under the Curve AUC(INF)
Description: Area under the serum concentration-time curve from time zero extrapolated to infinity
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
ug*h/mL | 35693.8 (22) | 38254.6 (16)
Statistical Analysis 1: Comparison: Cohort A (New Process) vs Cohort B (Current Process); Test type: Equivalence — Equivalence is concluded if the 90% CIs for the ratios of geometric means are contained within 0.8 to 1.25; Ratio of Geometric Means = 0.929, 90% CI 2-sided [0.884 to 0.976] — Cohort A vs Cohort B

3. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Time of maximum observed serum concentration
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
Hours | 1.000 [0.47 to 24.00] | 1.000 [0.25 to 24.00]

4. Secondary Outcome: Area Under the Curve AUC(0-T)
Description: Area under the serum concentration-time curve from zero to the last time of the last quantifiable concentration
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
ug*h/mL | 34473.2 (22) | 36671.6 (16)
Statistical Analysis 1: Comparison: Cohort A (New Process) vs Cohort B (Current Process); Test type: Equivalence — Equivalence is concluded if the 90% CIs for the ratios of geometric means are contained within 0.8 to 1.25; Ratio of Geometric Means = 0.936, 90% CI 2-sided [0.891 to 0.983] — Cohort A vs Cohort B

5. Secondary Outcome: Area Under the Curve AUC(0-28)
Description: Area under the serum concentration-time curve from time zero to 28 days after dosing
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
ug*h/mL | 28597.9 (20) | 29765.7 (15)
Statistical Analysis 1: Comparison: Cohort A (New Process) vs Cohort B (Current Process); Test type: Equivalence — Equivalence is concluded if the 90% CIs for the ratios of geometric means are contained within 0.8 to 1.25; Ratio of Geometric Means = 0.957, 90% CI 2-sided [0.915 to 1.001] — Cohort A vs Cohort B

6. Secondary Outcome: Total Body Clearance (CLT)
Description: Total body clearance
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/Kg
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
mL/h/Kg | 0.2642 (21) | 0.2445 (17)

7. Secondary Outcome: Volume of Distribution at Steady-State (Vss)
Description: Volume of distribution at steady-state
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/Kg
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
L/Kg | 0.10444 (21) | 0.10462 (21)

8. Secondary Outcome: Terminal Phase Elimination Half-life (T-HALF)
Description: Terminal phase elimination half-life in serum
Time Frame: From drug administration to 70 days following drug administration
Population: All treated participants with available concentration-time data
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 69 | 70
Hours | 357.464 (78.6519) | 369.425 (76.0162)

9. Secondary Outcome: Number of Participants Experiencing Positive Immunogenicity Response to Abatacept
Description: Positive immunogenicity response to Abatacept was defined if one of the following criteria was met:
  1. missing baseline immunogenicity measurement and a positive, post-baseline, laboratory-reported immunogenicity response;
  2. a negative laboratory-reported baseline immunogenicity response and a positive, post-baseline, laboratory-reported response;
  3. a positive, laboratory-reported, baseline immunogenicity response and a positive, post-baseline, laboratory-reported immunogenicity response with a titer value greater than the baseline titer value.
Time Frame: From Day 1 (Predose) to Day 71 (Study Discharge), assessed at day 1, day 29, day 57 and day 71
Population: All treated participants with available concentration-time data
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 70 | 70
Participants | 14 | 11

10. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing different types of Adverse Events (AEs). Peri-infusional AEs: occurring during the 30 minute study drug infusion period Post-infusional AEs: occurring within 24 hours post drug infusion
Time Frame: From drug administration to 56 days following drug administration
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 70 | 70
Participants
  Participants with at least 1 Adverse Event | 20 | 18
  Participants with at least 1 peri-infusional Adverse Event | 1 | 2
  Participants with at least 1 post-infusional Adverse Event | 4 | 3
  Participants with Adverse Event related to study drug | 8 | 7
  Death | 0 | 0
  Serious Adverse Events (SAEs) | 0 | 0
  Adverse Events leading to discontinuation | 0 | 0

11. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Mean Change from Baseline in systolic and diastolic blood pressure values
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
mmHg
  Systolic Blood Pressure | -0.3 (12.21) | 2.0 (10.72)
  Diastolic Blood Pressure | -0.8 (7.69) | -0.7 (8.52)

12. Secondary Outcome: Change From Baseline in Heart Rate
Description: Mean Change from Baseline in heart rate values
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
bpm | 1.6 (9.99) | 0 (9.34)

13. Secondary Outcome: Change From Baseline in Respiration Rate
Description: Mean Change from Baseline in respiration rate values
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: breath/min
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
breath/min | 1.0 (3.27) | 0.5 (3.63)

14. Secondary Outcome: Change From Baseline in Body Temperature
Description: Mean Change from Baseline in body temperature values
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: C
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
C | -0.01 (0.486) | -0.06 (0.392)

15. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Description: Mean Change from Baseline in ECG parameters, including PR interval, QRS interval, QT interval, and QTC Fridericia
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
msec
  PR Interval | 1.6 (17.66) | -1.8 (10.49)
  QRS Interval | 1.6 (5.70) | -0.0 (5.45)
  QT Interval | -1.1 (22.53) | -2.1 (17.28)
  QTC Fridericia | 1.4 (13.20) | 0.5 (12.70)

16. Secondary Outcome: Number of Participants Experiencing Clinically Significant Physical Examination Abnormalities
Description: Number of participants experiencing clinically significant physical examination abnormal findings
Time Frame: From the pre-treatment period to 70 days after start of study medication (approximately 100 days)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 70 | 70
Participants | 0 | 0

17. Secondary Outcome: Change From Baseline in Laboratory Test Results - Hematology 1
Description: Mean Change from Baseline in laboratory test results - Hematology parameters 1
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: x10*9 cells/L
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
x10*9 cells/L
  Platelet Count | 3.9 (30.99) | -1.6 (31.81)
  Basophils (absolute) | -0.026 (0.0741) | -0.015 (0.0292)
  Eosinophils (absolute) | -0.006 (0.1006) | 0.012 (0.012)
  Leukocytes | 0.09 (1.154) | -0.07 (1.225)
  Lymphocytes (absolute) | 0.073 (0.5086) | -0.028 (0.3162)
  Monocytes (absolute) | -0.045 (0.1163) | -0.033 (0.1453)
  Neutrophils (absolute) | 0.083 (0.9523) | -0.011 (1.0654)

18. Secondary Outcome: Change From Baseline in Laboratory Test Results - Hematology 2
Description: Mean Change from Baseline in laboratory test results - Hematology parameters 2
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
Fraction
  Basophils (relative) | -0.0034 (0.00779) | -0.0023 (0.00462)
  Eosinophils (relative) | -0.0008 (0.01712) | 0.0024 (0.01372)
  Lymphocytes (relative) | 0.0107 (0.07609) | 0.0019 (0.06250)
  Monocytes (relative) | -0.0073 (0.01389) | -0.0041 (0.02072)
  Neutrophils (relative) | 0.0008 (0.08609) | 0.0021 (0.07425)

19. Secondary Outcome: Change From Baseline in Laboratory Test Results - Hematology 3
Description: Mean Change from Baseline in laboratory test results - Hematocrit
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: Proportion of Blood Volume
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
Proportion of Blood Volume | -0.0017 (0.01845) | 0.0014 (0.01767)

20. Secondary Outcome: Change From Baseline in Laboratory Test Results - Chemistry 1
Description: Mean Change from Baseline in laboratory test results - Chemistry parameters 1
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
U/L
  Alanine Aminotransferase (ALT) | 0.6 (9.01) | -1.3 (8.50)
  Alkaline Phosphatase (ALP) | -3.0 (7.52) | -0.4 (8.86)
  Aspartate Aminotransferase (AST) | 1.1 (15.89) | -1.1 (4.11)
  Lactate Dehydrogenase (LD) | 1.4 (47.60) | -3.2 (18.30)

21. Secondary Outcome: Change From Baseline in Laboratory Test Results - Chemistry 2
Description: Mean Change from Baseline in laboratory test results - Chemistry parameters 2
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
umol/L
  Bilirubin, Direct | -0.01 (0.804) | -0.09 (0.759)
  Bilirubin, Total | -0.25 (3.467) | -0.54 (3.297)
  Creatinine | -2.2 (9.72) | -1.5 (8.58)

22. Secondary Outcome: Change From Baseline in Laboratory Test Results - Chemistry 3
Description: Mean Change from Baseline in laboratory test results - Chemistry parameters 3
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
mmol/L
  Blood Urea Nitrogen | 0.29 (1.264) | 0.12 (1.125)
  Calcium, Total | -0.027 (0.0809) | -0.012 (0.0787)
  Chloride, Serum | 0.4 (1.83) | -0.1 (2.01)
  Magnesium, Serum | -0.011 (0.0610) | -0.015 (0.0666)
  Phosphorus, Inorganic | -0.010 (0.1537) | -0.040 (0.1431)
  Potassium, Serum | -0.13 (0.266) | -0.23 (0.311)
  Sodium, Serum | -0.1 (2.22) | -0.2 (2.09)
  Glucose, Serum | 0.04 (0.516) | 0.04 (0.383)
  Uric Acid | 0.006 (0.0425) | 0.004 (0.0341)

23. Secondary Outcome: Change From Baseline in Laboratory Test Results -Hematology and Chemistry 4
Description: Mean Change from Baseline in laboratory test results - hematology and chemistry parameters 4
Time Frame: From baseline (last result before start of study medication) to 70 days after start of study medication
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
Number analyzed (Participants) | 67 | 67
g/L
  Hemoglobin (g/L) | -0.6 (6.06) | 0.4 (5.57)
  Albumin (g/L) | -0.9 (2.53) | -0.3 (2.39)
  Protein, Total (g/L) | -1.2 (4.50) | -0.4 (4.32)

ADVERSE EVENTS:
Time Frame: From drug administration to 70 days following drug administration
Arm/Group | Cohort A (New Process) | Cohort B (Current Process)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 6/70 | 3/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (New Process) (N=70) | Cohort B (Current Process) (N=70)
Nasopharyngitis (Infections and infestations) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03714022/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03714022/SAP_001.pdf